CLINICAL TRIAL: NCT05748873
Title: A Phase I/II Study to Assess the Safety and Tolerability of a Single Subretinal Administration of SPVN06 Gene Therapy in Subjects With Rod-Cone Dystrophy (RCD) Due to a Mutation in the RHO, PDE6A, or PDE6B Gene
Brief Title: Promising ROd-cone DYstrophy Gene therapY
Acronym: PRODYGY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SparingVision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPVN06-CLIN-01
Record Dates: First submitted 2023-02-07; First posted 2023-03-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-09

CONDITIONS: Retinitis Pigmentosa
Keywords: RHO; PDE6A; PDE6B; Pathogenic Mutation; Retinal Disease; Eye Disease; Rod-Cone Dystrophy; Gene Therapy; Retinal Dystrophies; Retinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Eye Diseases; Cone-Rod Dystrophies; Retinal Dystrophies; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Phase I/II study including an open-label dose-escalation phase (Step 1) and a three-arm, controlled, double-masked, randomized extension phase (Step 2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase I/II study including an open-label dose-escalation phase (Step 1) and a three-arm, controlled, double-masked, randomized extension phase (Step 2). In Cohorts 5 and 6 of Step 2, subjects and the designated study personnel will be masked to subject's dose assignment. Cohort 4 (untreated group) will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Step 1 : SPVN06 dose 1 (Experimental): Participants will receive a single subretinal injection of SPVN06 Dose 1 on Day 0.
  Interventions: Drug: SPVN06
- Step 1 : SPVN06 dose 2 (Experimental): Participants will receive a single subretinal injection of SPVN06 Dose 2 on Day 0
  Interventions: Drug: SPVN06
- Step 1 : SPVN06 dose 3 (Experimental): Participants will receive a single subretinal injection of SPVN06 Dose 3 on Day 0
  Interventions: Drug: SPVN06
- Step 2 : SPVN06 Dose Recommended 1 (Experimental): Participants will receive a single subretinal injection of SPVN06 recommended dose 1 on Day 0
  Interventions: Drug: SPVN06
- Step 2 : SPVN06 Dose Recommended 2 (Experimental): Participants will receive a single subretinal injection of SPVN06 recommended dose 2 on Day 0
  Interventions: Drug: SPVN06
- Step 2 : Control group (No Intervention)

INTERVENTIONS:
Drug: SPVN06 — AAV-RdCVF-RdCVFL
  Arms: Step 1 : SPVN06 dose 1; Step 1 : SPVN06 dose 2; Step 1 : SPVN06 dose 3; Step 2 : SPVN06 Dose Recommended 1; Step 2 : SPVN06 Dose Recommended 2

SUMMARY:
This is a two-step, multicenter, Phase I/II study including an open-label dose-escalation phase (Step 1) and a three-arm, controlled, double-masked, randomized extension phase (Step 2), in subjects with advanced RCD due to a mutation in the RHO, PDE6A, or PDE6B gene.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in this study only if all the following criteria apply:

1. Able to give signed informed consent and comply with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
2. Age ≥18 years at the time of ICF signature.
3. Subjects of either gender previously diagnosed with advanced RCD due to biallelic mutations in the rod cGMP phosphodiesterase 6 beta (PDE6B) or rod cGMP phosphodiesterase alpha (PDE6A) genes, or due to a monoallelic dominant mutation in the rhodopsin (RHO) gene. The genotyping results must be documented before the initiation of the Screening Visit. Subjects should be retested by the investigator if their genotyping tests were not performed within the 7 previous years, or if they were not performed by an accredited laboratory. In this case, the screening period can be prolonged for 2 additional weeks to allow time to generate genotyping results.
4. Advanced stage is defined as a stage of the natural history of the disease where both distance visual acuity and visual field are affected in both eyes. Substages within the advanced stage are defined as follows (monocular measurements, horizontal axis of isopter III4e for the visual field):

   * Severe stage is defined by both a BCVA below or equal to 20/200 and above or equal to 20/800, and a visual field below or equal to 20 degrees (subjects of Cohorts 1 to 3)
   * Intermediate stage is defined by both a BCVA below or equal to 20/40 and above 20/200, and a visual field below or equal to 20 degrees (subjects of Cohorts 4 to 6)
5. For subjects with severe advanced RCD enrolled in Step 1 only, the difference in visual acuity between the two eyes of a given subject should be equal to or below 0.3 logarithm of the minimal angle (LogMAR) (≤3 ETDRS lines), with a tolerance margin of 3 ETDRS letters.
6. Clinical diagnosis of RCD based on past medical and family history, mid-peripheral visual field dysfunction, photopsia, night blindness (nyctalopia), and fundoscopic appearance (including but not restricted to bone spicule pigmentation, attenuation of the retinal vessels, and waxy pallor of the optic nerve).
7. Diagnosis of RCD is confirmed on prior full-field ERG (any previously performed ERG is acceptable).
8. Documented preservation of cone inner and outer segments considered good enough by the investigator for the subject to be included in the study.
9. Negative serum pregnancy test for women of childbearing potential (please refer to Schedule of Assessments for details).
10. Women of childbearing potential (WOCBP) and men and/or their partner(s) of childbearing potential must agree to use a highly effective contraceptive method. This applies to the time period between ICF signature and 12 months after SPVN06 subretinal injection SRI (i.e., no longer applicable to subjects of Cohort 4 after randomization). The definition of highly effective contraceptive methods follows CTFG recommendations. Highly effective contraceptive methods are limited to:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

      * Oral
      * Intravaginal
      * Transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation:

      * Oral
      * Injectable
      * Implantable
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Sexual abstinence
11. Subjects must be affiliated to a health security system, if they are included in a clinical site based in France (per law).
12. No out-of-range values for clinical laboratory tests, however, if outside, must be considered as non-clinically relevant by the investigator using a multidisciplinary approach and compatible with a participation in the clinical study.
13. 12-lead electrocardiogram within normal limits, however, when outside, must be documented by the investigator using a multidisciplinary approach as not clinically relevant and compatible with a participation in the clinical study. Nota bene: This criterion of eligibility is only applicable to subjects assigned to a treatment cohort (Cohorts 1, 2, 3, 5, or 6), and is not required to authorize randomization in Step 2.
14. Physical examination without any clinical findings of clinical relevance (per medical/anesthesia staffs judgment) that could compromise participation in the clinical study or could affect the collection and/or evaluation of the study parameters. The findings of clinical relevance considered as contraindications to SPVN06 treatment include, but are not limited to, pulmonary pathology such as COPD, asthma, cardiac conditions such as congestive heart failure or valve disease, renal issues such as renal insufficiency and endocrine issues such as diabetes.

Exclusion Criteria:

Subjects are not eligible to participate in this study if any of the following criteria apply:

1. Subjects with prior administration of any gene therapy or any previous treatment with stem cell therapy for ocular or non-ocular disease.
2. Subjects participating in another clinical trial and receiving an investigational medicinal product (IMP) within 5 half-lives or 90 days prior to the injection of SPVN06.
3. Subjects with RCD due to any mutation in genes other than those listed in the inclusion criteria.
4. Subjects with systemic disease or other pathology not related to their diagnosis of RCD, and whose symptoms or associated treatments may affect vision, for example cancers or pathology of the central nervous system.
5. Subjects with narrow irido-corneal angles or any other medical situation contraindicating pupillary dilation.
6. Subjects known to be allergic to any of the delivery vehicle constituents or to any other drugs planned to be used during the clinical study.
7. Subjects with known allergies to corticosteroids, or who will be unable to tolerate the corticosteroid regimen as described in the protocol
8. Subjects with systemic disease or other medical or psychiatric conditions that preclude safe participation in the study.
9. Subjects receiving immunosuppressive therapies, other than the immune modulating regimen described in this protocol, or any other therapy known to influence the immune system including but not limited to steroid implants, cytostatics, interferons, tumor necrosis factor (TNF)-binding proteins, drugs acting on immunophilins, or antibodies with known impact on the immune system.
10. Subjects of reproductive potential unwilling to use effective contraception starting right after ICF signature and for 12 months after SPVN06 SRI (i.e., no longer applicable to subjects of Cohort 4 after randomization).
11. Subjects who are pregnant or breastfeeding.
12. Subjects who are unwilling or unable (based on the investigator's judgment) to comply with the study protocol.
13. Subjects with any condition that would not allow them to complete follow-up examinations during the study and, in the opinion of the investigator, would make them unsuitable for the study.
14. Subjects positive for human immunodeficiency virus (HIV) or any other systemic immunocompromising disease.
15. Subjects who have undergone, within 6 months before inclusion, any significant ocular surgery (per investigator's judgment) that could interfere with the evaluation of SPVN06 study objectives.
16. Presence of eye disorders that could interfere with the assessment of visual acuity and/or any other ocular assessments, including SD-OCT, during the study.
17. Presence of any systemic or ocular diseases, other than non-syndromic retinitis pigmentosa (RP), that can cause vision loss.
18. Prior vitrectomy or vitreomacular surgery.
19. Presence of vitreomacular adhesion or traction, epiretinal membrane macular pucker or macular hole, evident by ophthalmoscopy and/or SD-OCT examinations and assessed by the investigator to significantly affect central vision.
20. Current evidence of retinal detachment assessed by the investigator to significantly affect central vision.
21. Active ocular inflammation or recurrent history of idiopathic or autoimmune-associated uveitis.
22. Subjects with presence of any suspected or active ocular or periocular infection (conjunctivitis, keratitis, scleritis, endophthalmitis).
23. Subjects with history of glaucoma.
24. Subjects with uncontrolled intraocular pressure (IOP).
25. Subjects with active cancer or currently receiving any therapy for cancer treatment.
26. Subjects with any history of ocular malignancy.
27. Subjects with a clinically significant cardiac disease on routine clinical examination (history, physical examination), or known congestive heart failure, myocardial infarction, clinically significant valvular heart disease, clinically significant cardiac rhythm or conduction abnormalities.
28. Subjects with unstable/uncontrolled hypertension, defined by national recommendations.
29. Subjects with pulmonary dysfunction or severe obstructive pulmonary disease.
30. Subjects with active tuberculosis.
31. Subjects with liver or renal insufficiency.
32. Subjects with unstable endocrine disease, including unstable diabetes or thyroid disease.
33. Subjects with active Hepatitis B or Hepatitis C.
34. Subjects with clinically active infection of herpetic diseases, including herpes simplex virus, varicella zoster virus (VZV), cytomegalovirus (CMV) or EBV.
35. Subjects with known history of ocular infection with herpes simplex virus.
36. Subjects with active (extraocular) infection (requiring or not the prolonged or chronic use of antimicrobial agents).
37. Immunocompromised subjects with previous solid organ or bone marrow transplant.
38. Subjects who receive a live vaccine less than 4 weeks prior to SPVN06 injection
39. Subjects who were infected by COVID-19 less than 2 weeks prior to SPVN06 injection.
40. Subjects who have recently received (less than 4 weeks) or plan to receive a COVID-19 vaccination.
41. Incapacitated subjects, as defined by national laws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of a single injection of SPVN06 in subjects with advanced RCD due to a mutation in the RHO, PDE6A, or PDE6B gene, 12 months after administration of gene therapy. | Baseline to 12 months after administration of gene therapy
  Incidence and severity of systemic and ocular AEs and SAEs

SECONDARY OUTCOMES:
Evaluation of the long-term safety and tolerability of a single injection of SPVN06 in subjects with advanced RCD due to a mutation in the RHO, PDE6A, or PDE6B gene, up to 5 years after treatment administration. | up to 5 years after treatment
  Incidence and severity of systemic and ocular AEs and SAEs
Evaluation of viral shedding and bio-dissemination up to 1 year after treatment administration. | up to 1 year after treatment
  Quantification of viral DNA copies in tears (viral shedding) and in blood (bio-dissemination)
Evaluation of the immune response against the viral vector and the transgene products of SPVN06 up to 5 years after treatment administration. | up to 5 years after treatment
  Titration of total antibodies against the viral capsid
Evaluation of preliminary efficacy as assessed by visual acuity | up to 5 years after treatment
  BCVA change from baseline (EDTRS chart)
Evaluation of preliminary efficacy as assessed by optical coherence tomography | up to 5 years after treatment
  Anatomical change from baseline (SD-OCT)
Evaluation of preliminary efficacy as assessed by color vision | up to 5 years after treatment
  Change from baseline of parameters collected by color vision assessment
Evaluation of preliminary efficacy as assessed by visual field | up to 5 years after treatment
  Change from baseline of static perimetry, kinetic perimetry and microperimetry
Evaluation of preliminary efficacy as assessed by retinal sensitivity | up to 5 years after treatment
  Change from baseline of parameters collected by full-field electroretinography
Evaluation of preliminary efficacy as assessed by retinal sensitivity | up to 5 years after treatment
  Change from baseline of parameters collected by FST
Evaluation of preliminary efficacy as assessed by FAF | up to 5 years after treatment
  Change from baseline of parameters collected by fundus autofluorescence
Evaluation of preliminary efficacy as assessed by quality of life | up to 5 years after treatment
  Change from baseline of parameters collected by VFQ-25
Evaluation of preliminary efficacy as assessed by quality of life | up to 5 years after treatment
  Change from baseline of parameters collected by ViSIO-PRO

OTHER OUTCOMES:
Exploratory objective - Exploration of biomarkers | up to 5 years after treatment
  Collect and store urine and blood (in addition to the body fluids used for the assessment of viral shedding and bio-dissemination) for further exploration of biomarkers of medical interest not already identified at time of protocol submission.
Exploratory objective - Photoreceptor mosaic imaging | up to 5 years after treatment
  Collect and analyze photoreceptor mosaic images using adaptive optics

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Bascom Palmer Eye Institute/University of Miami, Miami, Florida
  - Mass Eye and Ear, Boston, Massachusetts
  - Casey Eye Institute, Portland, Oregon
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
- CHNO XV-XX Paris - CIC 1423, Paris, France

REFERENCES:
- [Derived] Marie M, Churet L, Gautron AS, Farjo R, Mizuyoshi K, Stevenson V, Khabou H, Leveillard T, Sahel JA, Lorget F. Preclinical safety and biodistribution of SPVN06, a novel gene- and mutation-independent gene therapy for rod-cone dystrophies. Gene Ther. 2025 Aug 4. doi: 10.1038/s41434-025-00556-3. Online ahead of print. PMID 40759732